CLINICAL TRIAL: NCT02842684
Title: Orthopedic Digital Planning for Total Hip Arthroplasties
Acronym: ORTHOPLAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/14/7426
Record Dates: First submitted 2016-07-20; First posted 2016-07-25 (Estimated); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Infection of Total Hip Joint Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traumacad software (Experimental): Preoperative planning of hip prothesis is practiced by layer on radiographs whose scaling is imprecise . The recent TraumaCad system ( Brainlab® ) allows adjustment of the scales for each patient and the virtual positioning of implants to simulate the response to the return of geometric hip parameters
  Interventions: Device: TraumaCad software
- without digital planning (No Intervention): Preoperative planning of hip prothesis is practiced by layer on radiographs whose scaling is imprecise

INTERVENTIONS:
Device: TraumaCad software — restitution of anatomical- radiological parameters after total hip arthroplasty with TraumaCad , conventional planning systems and without planning.
  Arms: Traumacad software

SUMMARY:
Preoperative planning has been carried out to allow for response preparedness . A layer technique is usually used with standard radiography .The investigators have a record of routine preoperative radiographs by standard recognized as having an advantage over the reproducibility of measurements compared with plain radiography . The Toulouse Hospitals have developed this technology and is part of the routine assessment of hip prothesis pre and postoperatively.

The TraumaCad software can superimpose implants on Picture Archiving and Communication System and evaluate digital and reproducible size of the implants and their correct position .

This is to demonstrate the superiority of modern digital tools in the preoperative preparation in Orthopaedics set.

DETAILED DESCRIPTION:
Modern joint replacements in orthopedic surgery allow to restore locomotion. More than 150,000 hip replacements are performed each year in France . The optimization results going restoration of the lengths of members and anatomy .

Preoperative planning of hip replacements optimizes the return of the hip rotation center . Preoperative planning of hip prothesis is practiced by layer on radiographs whose scaling is imprecise . The recent TraumaCad system ( Brainlab® ) allows adjustment of the scales for each patient and the virtual positioning of implants to simulate the response to the return of geometric parameters of the hip.

Preoperative planning by TraumaCad hip arthroplasties provides better restitution of limb length over conventional planning methods.

The standardized radiographs being the investigators want to compare this group with a control group operated without TraumaCad planning and evaluating the accuracy of the software to predict implants sizes also .

There is no risk to the patient with this procedure . The direct benefit is increased accuracy of surgical gesture to the patient and the reduction of mechanical problems related to leg length . Earnings for the orthopedic community is the postoperative evaluation. In the long term , the prosthetic technical improvement must increase the life of prostheses with therefore lower revisions and less expenditure in terms of public health.

The widespread use of automated planning and objective assessment postoperative radiographs .

ELIGIBILITY:
Inclusion Criteria:

* Inclusion concerns all major patients able supported for osteoarthritis for the realization of a primary hip replacement .

Exclusion Criteria:

* Minor patients
* BMI greater than 35 patients
* Recovery or major architectural disorder surgery ( preoperative upper inequality 2 cm or dysplastic hip)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
postoperative inequality measured on the radiograph the 3rd postoperative day. | day 3 after chirurgical intervention
  postoperative inequality measured on the radiograph the 3rd postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Reina, Dr, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No